CLINICAL TRIAL: NCT00037947
Title: Auditory Function in Patients With and Without Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2568R
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Hearing
MeSH Terms: conditions — Multiple Sclerosis | interventions — Hearing

INTERVENTIONS:
Procedure: Hearing in Multiple Sclerosis

SUMMARY:
We propose to evaluate auditory function and neuropsychologic function in 150 Multiple Sclerosis (MS) patients and in 150 patients who do not have MS. Experimental subjects will be recruited by selecting patients with a verified diagnosis of MS from the registry of patients established by the Oregon Health Sciences University, Multiple Sclerosis Research Center. Control subjects will be matched with respect to age, to gender and to audiometric configuration.

DETAILED DESCRIPTION:
This study will compare the prevalence and nature of hearing dysfunction in patients with MS and in a group of control subjects without MS. The work will address three main goals:

1. Evaluating the possibility that MS is a risk factor for hearing impairment, tinnitus and central auditory dysfunction.
2. Determining the nature and the extent of auditory dysfunction in individuals with MS compared to those without MS; and determining neuropsychological function in each group.
3. Evaluating the extent to which disability in individuals with MS may be amplified by the presence of auditory dysfunction.

Measurements of auditory function and psychometric performance will be compared between MS patients and control subjects without MS. These subjects will come to the Portland VAMC for four sessions of comprehensive auditory and psychometric testing. Additional information on disease history and status, hearing history, and current-disability status will be obtained.

Subjects The patient group (Group 1) will consist of 150 patients with diagnosed MS, recruited at the MS Center of Oregon. For this group, inclusion criteria for each patient will include: (1) a clinical or laboratory supported diagnosis of "definite MS" (Poser, et al., 1983); (2) a diagnosis of relapsing, remitting or secondary progressive MS; (3) A Kurtzke Expanded Disability Status Score (EDSS) of 0 to 7.0, inclusive; (4) no history of a clinical relapse or change in EDSS for three months preceding entry into the study; and (5) a brain MRI scan (within the preceding year) that shows at least three white-matter lesions on T2-weighted images consistent with MS.

The control group (Group 2) will consist of 150 subjects without MS who are matched to the patient group with respect to age (± 5 years), to gender and to audiometric configuration (within ±10 dB Hearing Level for the octave test frequencies from 500 through 8000 Hz). Subjects in Group 2 will be recruited from the VA audiology clinic and from a cohort of more than 360 subjects and patients who have been used as controls in five other studies. Both males and non-pregnant females will be recruited in equal numbers. Minority individuals will be recruited in accordance with recommendations for proportional minority representation established by the Office of Human Research Accountability and the Minority Affairs Program. The protocols will be explained verbally by the investigators, and restated in consent forms approved by the VA IRB, and signed by the subject, by the investigator and by a witness.

ELIGIBILITY:
Multiple Sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2001-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wolff, Ph.D. Special Assistant to the Director — Program Analysis and Review Section (PARS), VA Rehabilitation Research & Development Service; Danielle Kerkovitch, Ph.D. — Program Analysis and Review Section (PARS), VA Rehabilitation Research and Development Service
Locations (1):
- VA Medical Center, Portland, Oregon, United States